CLINICAL TRIAL: NCT06229314
Title: Effect of Inspiratory Muscle Training on Respiratory Function, Exercise Capacity, and Quality of Life in Operated Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial
Brief Title: Effect of Inspiratory Muscle Training in Operated Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Ukbe Sirayder, Principal Investigator, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/165
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Scoliosis Idiopathic Adolescent

STUDY DESIGN:
Intervention Model Description: In this study, the preoperative pulmonary function, respiratory and peripheral muscle strengths, functional capacities, and QoL of AIS patients who were eligible for surgery by the physician were evaluated. Subsequently, individuals underwent surgery. Pulmonary function tests and respiratory muscle strength measurements were performed on the patients approximately two days after surgery. Inspiratory Muscle Training was initiated at 60% of the MIP value. IMT was administered using the Powerbreathe device twice a day with 30x2 breaths. The device was adjusted weekly based on the patient's current MIP value, and training continued at 60% of the MIP value . The sham group received IMT at 5% of the measured MIP value, with adjustments made weekly, similar to the IMT group. Patients were asked to keep a daily record of their sessions. IMT was administered for a total of 6 weeks. At the end of the sixth week, initial tests and questionnaires were repeated for individuals in both groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT Group (Experimental): The IMT group received IMT at 60% of the measured MIP value. IMT was administered using the Powerbreathe device (Powerbreathe Plus, Warwickshire, England) twice a day with 30x2 breaths. The device was adjusted weekly based on the patient's current MIP value, and training continued at 60% of the MIP value.
  Interventions: Device: Inspiratory muscle training
- Control Group (Sham Comparator): The sham group received IMT at 5% of the measured MIP value, with adjustments made weekly, similar to the IMT group. Patients were asked to keep a daily record of their sessions. IMT was administered for a total of 6 weeks.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — In this study, the preoperative pulmonary function, respiratory and peripheral muscle strengths, functional capacities, and QoL of AIS patients who were eligible for surgery by the physician were evaluated. Subsequently, individuals underwent surgery. Pulmonary function tests and respiratory muscle strength measurements were performed on the patients approximately two days after surgery. Inspiratory Muscle Training was initiated at 60% of the MIP value. IMT was administered using the Powerbreathe device twice a day with 30x2 breaths. The device was adjusted weekly based on the patient's current MIP value, and training continued at 60% of the MIP value . The sham group received IMT at 5% of the measured MIP value, with adjustments made weekly, similar to the IMT group. Patients were asked to keep a daily record of their sessions. IMT was administered for a total of 6 weeks. At the end of the sixth week, initial tests and questionnaires were repeated for individuals in both groups.

SUMMARY:
In adolescent idiopathic scoliosis (AIS), if the appropriate treatment approach is not applied, the patient's general health condition is negatively affected by the deterioration of pulmonary function. Although studies in the literature evaluate individuals with AIS and investigate the effects of exercise training on their functional capacity, no study has been found examining the effectiveness of post-surgical respiratory muscle strength training (IMT). Therefore, this study was designed as a randomized controlled study with the aim of investigating the effectiveness of IMT in the early post-surgical period in individuals with AIS. Participants included individuals diagnosed with AIS, for whom a surgical decision was made by an orthopedic surgeon, and who could cooperate in the tests to be conducted. Twelve patients were in the IMT group, and 12 were in the sham group. Pulmonary function and respiratory and peripheral muscle strength were measured. Functional capacities were assessed using the Six-Minute Walk Test (6MWT). Disease-specific quality of life (QoL) was evaluated through the Scoliosis Research Society-22 (SRS-22) and Oswestry Low Back Pain Questionnaire, while dyspnea was assessed using the Modified Medical Research Council (mMRC) scale. In the IMT group, IMT was provided at 60% of the Maximum Inspiratory Pressure (MIP), while in the Sham group, IMT was provided at 5% of MIP.

DETAILED DESCRIPTION:
There are very few studies in the literature that have investigated the effects of Inspiratory Muscle Training (IMT) to individuals with scoliosis. In a study conducted by Kim et al. in 2005, individuals with scoliosis and spinal cord injuries were given IMT, and after treatment, a decrease in Cobb angles, a significant increase in lung volumes, and respiratory muscle strengths were observed. In a study by Basbug et al. in 2023, the impact of IMT on pulmonary function and functional capacity in individuals with AIS was investigated. There is no study in the literature on providing IMT after surgery in scoliosis patients. It has been shown that surgical treatment alone in scoliosis patients is insufficient to improve respiratory capacity in the short term. Therefore, in this study, we aimed to investigate the effects of postoperative IMT on pulmonary function, functional capacity, and quality of life in AIS patients.

Methods Trial design

This study was planned as a single-blind, randomized, parallel group clinical trial. Participants did not know which group they were in.

Participants

Patients admitted to Kayseri System Hospital between February 2023 and December 2023 and diagnosed with idiopathic scoliosis were included in the study. Data were collected at Nuh Naci Yazgan University Department of Physiotherapy and Rehabilitation Laboratories. We calculated (G*Power Version 3.1.9.4, Franz Faul, Universitat Kiel, Düsseldorf, Germany) a power of 80% with 0.05 significance, a difference to be detected of 0.84 liter, and a standard deviation of 0.59 liter in FVC value, generating a sample of 10 individuals per group. It was planned to take a total of 24 individuals, 12 individuals in each group, by calculating a minimum 20% drop-out rate. A total of 24 individuals, 12 in the IMT group and 12 in the sham group were included in the study.

The study included voluntary individuals diagnosed with AIS, who had been determined eligible for surgery by an orthopedic specialist, were able to cooperate in the tests, and did not have any orthopedic, cardiac, pulmonary, vestibular or neurological diseases other than scoliosis. Participants who had experienced acute infections within the last 15 days were excluded. The data were collected from February 2023 to December 2023.

Randomization

Twenty-four individuals were randomly selected using the computerized randomization method (www.random.org, Dublin, Ireland) among 29 individuals who met the inclusion criteria and volunteered to participate in the study. Then, two numbers series of 12 randomly prepared numbers with numbers between 1 and 24 were created using the computerized randomization method. Based on randomization, the group consisting of the first number series was accepted as the exercise group and the other as the control group. Afterward, the numbers from 1 to 24 were written on paper and put in 24 sealed envelopes. The patients in the study randomly chose an envelope when they came to their appointment and were included in the group where the number series with the chosen number coincided.

Materials

First, sociodemographic information of all individuals included in the study was obtained, and all questionnaires were conducted. Cobb angle was determined by the orthopedist using radiological imaging methods.

Dyspnea was evaluated using the Modified Medical Research Council (mMRC) dyspnea scale. It is a categorical scale in which individuals choose the most appropriate of the five expressions of dyspnea, between 0-4 points, to define their dyspnea levels.

A spirometer (Cosmed Pony FX Spirometer, Milan, Italy) was used to measure forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, peak expiratory flow rate (PEF), and forced expiratory volume from 25-75% (FEF25-75%), based on the European Respiratory Society/American Thoracic Society (ERS/ATS) criteria. The test was performed in the sitting position. At least three technically acceptable measurements were obtained between the two best-measured FEV1 values, with no more than a 5% difference, and the best FEV1 value was selected for analysis.

Respiratory muscle strength was measured (Cosmed Pony FX Spirometer, Milan, Italy). For the measurement of maximum inspiratory pressure (MIP), maximum expiration was performed on the person, and the respiratory tract was immediately closed with a valve. Then, the person was asked to perform maximum inspiration for 1-3 sec. For maximum expiratory pressure (MEP), a maximal inspiration was performed, and then the person was asked to perform a maximal expiration of 2 sec against the closed airway. At least three technically acceptable maneuvers were performed, with no more than a 5% difference between the two best-measured values.

Peripheral muscle strength was determined by measuring handgrip and quadriceps muscle strength using a digital dynamometer (Jtech Commander Muscle Tester, UT, USA). The mean values of the right and left side measurements were obtained. Then, the average of the measurements of the right and left sides were recorded in Newton (N) using each side.

The functional capacity of individuals was evaluated using the Six-Minute Walk Test (6MWT). Before and after the 6MWT, heart rate, blood pressure, oxygen saturation (SpO2) (Cosmed Spiropalm 6MWT, Rome, Italy), and respiratory frequency were assessed, and fatigue levels during exertion and dyspnea were evaluated using the Modified Borg Scale.

The disease-specific QoL for the cases was assessed using the Scoliosis Research Society-22 (SRS-22) scale. The Turkish version of the scale was used. Additionally, the Oswestry questionnaire was used to assess how much back pain affected daily activities.

Intervention

In this study, the primary outcome measurement was the pulmonary function test, and the secondary outcome measurements were dyspnea, respiratory and peripheral muscle strength, functional capacity and QoL. In the preoperative period, dyspnea, pulmonary function, respiratory and peripheral muscle strength, and QoL were evaluated, respectively. Finally, functional capacity was measured with 6MWT. Subsequently, individuals underwent surgery. Pulmonary function tests and respiratory muscle strength measurements were performed on the patients approximately two days after surgery (post-op). Inspiratory Muscle Training (IMT) was initiated at 60% of the MIP value. IMT was administered using the Powerbreathe device (Powerbreathe Plus, Warwickshire, England) twice a day with 30x2 breaths. The device was adjusted weekly based on the patient's current MIP value, and training continued at 60% of the MIP value. The sham group received IMT at 5% of the measured MIP value, with adjustments made weekly, similar to the IMT group. Patients were asked to keep a daily record of their sessions. IMT was administered for a total of 6 weeks. At the end of the sixth week (post-op sixth week), initial tests and questionnaires were repeated for individuals in both groups.

ELIGIBILITY:
Inclusion Criteria:

* did not have any orthopedic, cardiac, pulmonary, vestibular or neurological diseases other than scoliosis.

Exclusion Criteria:

* had experienced acute infections within the last 15 days were excluded

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | Six week
  A spirometer (Cosmed Pony FX Spirometer, Milan, Italy) was used to measure forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, peak expiratory flow rate (PEF), and forced expiratory volume from 25-75% (FEF25-75%), based on the European Respiratory Society/American Thoracic Society (ERS/ATS) criteria. The test was performed in the sitting position. At least three technically acceptable measurements were obtained between the two best-measured FEV1 values, with no more than a 5% difference, and the best FEV1 value was selected for analysis.

SECONDARY OUTCOMES:
Dyspnea | Six week
  Dyspnea was evaluated using the Modified Medical Research Council (mMRC) dyspnea scale. It is a categorical scale in which individuals choose the most appropriate of the five expressions of dyspnea, between 0-4 points, to define their dyspnea levels
Respiratory muscle strength | Six week
  Evaluated using spirometry device
Peripheral muscle strength | Six week
  Evaluated using digital dynamometer
Functional capacity | Six week
  Six Minute Walk Test is used
Quality of Health | Six week
  Scoliosis Research Society-22 (SRS-22) scale. The scale consists of 22 questions and 5 question subgroups. Subgroups; It consists of pain, evaluation of general appearance, spinal functions, mental health and satisfaction with treatment. The score range of the scale is "0 - 110". Higher scores indicate more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ukbe ŞIRAYDER, Dr., Principal Investigator — Nuh Naci Yazgan University
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No